CLINICAL TRIAL: NCT00286351
Title: Use of Arimidex and Zoladex as Pretreatment to IVF in Women With Ovarian Endometriosis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: endo 220604
Record Dates: First submitted 2006-02-01; First posted 2006-02-03 (Estimated); Last update posted 2007-04-23 (Estimated); Status verified 2007-04

CONDITIONS: Endometriosis
MeSH Terms: conditions — Endometriosis | interventions — Combined Modality Therapy; Anastrozole

INTERVENTIONS:
Drug: Combined treatment with Arimidex and Zoladex before IVF

SUMMARY:
Does a combination of Arimidex and Zoladex make endometriomas shrink and how is the following IVF outcome

ELIGIBILITY:
Inclusion Criteria:

* Endometrioma(s)with a size of 20-70 mm, persisted for at least 3 cycles
* Couples with indication and wish for IVF/ICSI
* Age of women: 20-40 years
* Regular menstrual cycle within normal range (21-35 days)
* Body Mass Index (BMI): 18-30 kg/m2

Exclusion Criteria:

* History with osteoporosis, liver-, kidney- or heart disease or thromboembolic disease
* Treatment of endometriosis with GnRH agonist during the last 3 month

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20
Dates: Start 2005-01

PRIMARY OUTCOMES:
size of endometriomas after 2½ month of combined downregulation

CONTACTS AND LOCATIONS:
Overall Officials: Kristine Lossl, medical doctor, Principal Investigator — The Fertility Clinic, Copenhagen University Hospital Rigshospitalet
Locations (1):
- The Fertility Clinic, Copenhagen University Hospital, Rigshospitalet, Copenhagen, Copenhagen East, Denmark